CLINICAL TRIAL: NCT03199313
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Sutezolid in Healthy Adult Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Sutezolid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sutezolid - CL001
Record Dates: First submitted 2017-06-23; First posted 2017-06-26 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary
Keywords: tuberculosis; TB; Sutezolid; pulmonary tuberculosis
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary | interventions — PNU-100480

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort 1 Sentinel Group 1 - Active (Active Comparator): N = 2, Initial dosing of Cohort 1 with 300 mg sutezolid or matching placebo, dosed 24 hours before the rest of Cohort 1 Group 2
  Interventions: Drug: Sutezolid
- Cohort 1 Sentinel Group 1 - Placebo (Placebo Comparator): N = 1, Initial dosing of Cohort 1 with 300 mg sutezolid or matching placebo, dosed 24 hours before the rest of Cohort 1 Group 2
  Interventions: Drug: Placebo
- Cohort 1 Sentinel Group 2 - Active (Active Comparator): N = 4, Secondary dosing of Cohort 1 with 300 mg sutezolid or matching placebo, dosed 24 hours after the rest of Cohort 1 Group 1
  Interventions: Drug: Sutezolid
- Cohort 1 Sentinel Group 2 - Placebo (Placebo Comparator): N = 1, Secondary dosing of Cohort 1 with 300 mg sutezolid or matching placebo, dosed 24 hours after the rest of Cohort 1 Group 1
  Interventions: Drug: Placebo
- Cohort 2 - Active (Active Comparator): N = 6, 600mg sutezolid or matching placebo
  Interventions: Drug: Sutezolid
- Cohort 2 - Placebo (Placebo Comparator): N = 2, 600mg sutezolid or matching placebo
  Interventions: Drug: Placebo
- Cohort 3 - Active (Active Comparator): N = 6, 1200 mg sutezolid or matching placebo
  Interventions: Drug: Sutezolid
- Cohort 3 - Placebo (Placebo Comparator): N = 2, 1200 mg sutezolid or matching placebo
  Interventions: Drug: Placebo
- Cohort 4 - Active (Active Comparator): N = 6, 1800 mg sutezolid or matching placebo
  Interventions: Drug: Sutezolid
- Cohort 4 - Placebo (Placebo Comparator): N = 2, 1800 mg sutezolid or matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sutezolid — Sutezolid supplied as tablets and matching placebo for oral administration.
  Other Names: PNU-100480
  Arms: Cohort 1 Sentinel Group 1 - Active; Cohort 1 Sentinel Group 2 - Active; Cohort 2 - Active; Cohort 3 - Active; Cohort 4 - Active
Drug: Placebo — Matching Sutezolid placebo
  Other Names: Placebo Oral Tablet
  Arms: Cohort 1 Sentinel Group 1 - Placebo; Cohort 1 Sentinel Group 2 - Placebo; Cohort 2 - Placebo; Cohort 3 - Placebo; Cohort 4 - Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose study conducted at one study center in the United States. Four (4) cohorts of 8 subjects each (6 active and 2 placebo). Subjects will participate in only one cohort.

Safety will be assessed throughout the study; serial ECGs and serial blood samples will be collected for the safety and PK assessment of sutezolid.

Dose escalation to the next cohort (i.e., dose level) will not take place until the Sponsor, in conjunction with the Principal Investigator, has determined that adequate safety, tolerability and PK from the previous cohort has been demonstrated to permit proceeding to the next cohort.

Interim PK analyses will be performed for the dose escalation decisions to reconsider the sampling time points as the study progresses. All samples will be sent for analysis and the bioanalytical lab will be unblinded and only run the analysis on active treatment subjects. Data from the analysis used for the escalation meetings will only include active treatment subjects, and will be blinded by subject.

Subjects will be housed in the clinic from at least 24 hours prior (from Day -2), until 48 hours (Day 3) after dosing. Subjects will be contacted via a phone call for follow-up questioning about adverse events 7 days later (Study Day 10).

ELIGIBILITY:
Inclusion Criteria:

1. Subject understands study procedures and provides written, informed consent prior to all trial-related procedures.
2. Healthy adult male and females of non-childbearing potential, 19 to 50 years of age (inclusive) at the time of screening.
3. < Body mass index (BMI) ≥ 18.5 and ≤ 32.0 (kg/m2) and a body weight of no less than 50.0 kg.
4. Medically healthy with no clinically significant, as determined by the Investigator, screening results (e.g., laboratory profiles are normal or up to Grade 1 per Division of Microbiology and Infectious Diseases [DMID] Toxicity Tables) medical history, vital signs, ECGs, physical examination findings. Laboratory results within the testing facility's normal range will not be considered AEs when referenced to the DMID assessment/grading scale. If exclusionary laboratory criteria are met, values may be confirmed by repeat evaluation.
5. No use of tobacco or nicotine containing products (including smoking cessation products), for a minimum of 6 months prior to dosing.
6. Females of non-childbearing potential, having undergone one of the following sterilization procedures at least 6 months prior to dosing:

   1. Hysteroscopic sterilization
   2. Bilateral tubal ligation or bilateral salpingectomy
   3. Hysterectomy
   4. Bilateral oophorectomy
   5. or be postmenopausal with amenorrhea for at least 1 year prior to the first dose with serum follicle stimulating hormone (FSH) levels consistent with postmenopausal status at screening.
7. Non-vasectomized males (or males vasectomized less than 120 days prior to study start), must agree to the following during study participation and for 90 days following the last administration of study drug:

   1. use a condom with spermicide while engaging in sexual activity or be sexually abstinent
   2. not donate sperm during this time. In the event the sexual partner is surgically sterile, use of a condom with spermicide is not necessary. None of the restrictions listed above are required for vasectomized males whose procedure was performed more than 120 days prior to study start.

   In the event the sexual partner is surgically sterile, use of a condom with spermicide is not necessary. None of the restrictions listed above are required for vasectomized males whose procedure was performed more than 120 days prior to study start.
8. Willing to answer inclusion and exclusion criteria questionnaire at check-in.
9. Be able to comply with the protocol and the assessments therein, including all restrictions.
10. Is willing and able to remain in the study unit for the entire duration of the assigned confinement period and receive a phone call for follow-up questioning about AEs.

Exclusion Criteria:

Subjects will be excluded from the study if there is evidence of any of the following criteria at screening or check-in, as appropriate.

Medical History

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease as determined by the Investigator to be clinically relevant.
2. History of any illness that, in the opinion of the Investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
3. Surgery within the past 90 days prior to dosing as determined by the Investigator to be clinically relevant, or any history of cholecystectomy.
4. History or presence of alcoholism or drug abuse within the past 2 years as determined by the Investigator to be clinically relevant.
5. History of sensitivity or contraindication to use of linezolid or any study investigational products.
6. Female subjects who are pregnant or lactating.
7. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
8. Heart rate is lower than 40 bpm or higher than 99 bpm at screening.
9. Any clinically significant electrocardiogram abnormality at Screening (as deemed by decision of the Investigator and the Sponsor's Medical Monitor).

   NOTE: The following can be considered not clinically significant without consulting the Sponsor's Medical Monitor:
   1. Mild first degree A-V block (P-R interval <0.23 sec)
   2. Right or left axis deviation
   3. Incomplete right bundle branch block
   4. Isolated left anterior fascicular block (left anterior hemiblock) in younger athletic subjects
10. QTcF interval >450 msec for males or >470 msec for females at screening, Day -2, Day -1, or Day 1 (pre-dose), or history of prolonged QT syndrome.
11. Family history of Long-QT Syndrome or sudden death without a preceding diagnosis of a condition that could be causative of sudden death (such as known coronary artery disease, congestive heart failure or terminal cancer).
12. History of one or any combination of, the following:

    1. Seizures or seizure disorders
    2. Brain surgery.
    3. History of head injury in the last five years
    4. Any serious disorder of the CNS or related neurological system, particularly one that may lower the seizure threshold.
    5. History of seizures Specific Treatments
13. Use of any prescription medication within 14 days prior to dosing.
14. Use of any over-the-counter (OTC) medication, including herbal products and vitamins, within the 7 days prior to dosing, except acetaminophen. Up to 3 grams per day of acetaminophen is allowed at the discretion of the Investigator prior to dosing.
15. Use of any drugs or substances known to be significant inhibitors of Cytochrome P450 (CYP) enzymes and/or significant inhibitors or substrates of P-glycoprotein (P-gp) and/or Organic anion transporting polypeptides (OATP) within 14 days prior to the first dose of study drug.
16. Use of any drugs or substances known to be inducers of CYP enzymes and/or P-gp, including St. John's Wort, within 28 days prior to the first dose of study drug.
17. Use of any drugs or substance known to lower the seizure threshold.
18. Blood donation or significant blood loss within 56 days prior to dosing.
19. Plasma donation within 7 days prior to dosing.
20. Participation in another clinical trial within 28 days prior to dosing.
21. Consumption of the following prior to dosing period:

    1. Alcohol - 48 hours prior to dosing
    2. Grapefruit/Mandarin Oranges - 10 Days prior to dosing
    3. Caffeine/Xanthine - 24 hours prior to dosing Laboratory Abnormalities
22. Positive results for the urine drug/alcohol screen at screening or check-in.
23. Positive urine cotinine at screening.
24. Serum magnesium potassium, or calcium laboratory values outside of the normal range at screening. If exclusionary lab criteria are met, values may be confirmed by repeat evaluation.
25. Positive results at screening for Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HBsAg), or Hepatitis C antibodies (HCV).
26. Is unwilling to remove any artificial nails (e.g. acrylic, gel) or fingernail polish and not use such products for the duration of the study.
27. Is receiving any of the following medications: monoamine oxidase (MAO) inhibitors (phenelzine, tranylcypromine), tricyclic antidepressants (amitriptyline, nortriptyline, protriptyline, doxepin, amoxapine, etc.), antipsychotics such as chlorpromazine and buspirone, serotonin re-uptake inhibitors (fluoxetine, paroxetine, sertraline, etc.), buproprion, agents known to prolong the QTc interval (erythromycin, clarithromycin, astemizole, type Ia [quinidine, procainamide, disopyramide] and III [amiodarone, sotalol] anti-arrhythmics, carbamazepine, sulfonylureas, and meperidine), within 30 days before the first dose of study drug or during the study drug treatment period.
28. Use of any adrenergic/serotonergic agonists, such as pseudoephedrine and phenylpropanolamine (frequently found in cold and cough remedies), within 7 days before the first dose of study drug or during the study drug treatment period.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2017-12-16 (Actual); Study Completion 2017-12-16 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single oral doses of sutezolid in healthy adult subjects evaluated by Treatment Emergent Adverse Events (TEAEs) | Days 0-10
  Safety will be evaluated by Treatment Emergent Adverse Events (TEAEs) following doses of sutezolid or placebo

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of single oral doses of sutezolid using Cmax | Days 0-10
  This will be measured through PK parameters like Cmax; Cmax = maximum observed concentration
Pharmacokinetics (PK) of single oral doses of sutezolid using AUC | Days 0-10
  This will be measured through PK parameters like AUC; AUC = Area under the curve,
Pharmacokinetics (PK) of single oral doses of sutezolid using Tmax | Days 0-10
  This will be measured through PK parameters like Tmax; Tmax = Time of the maximum drug concentration (obtained without interpolation)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bruinenberg, MD, Study Director — Global Alliance for TB Drug Development
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States